CLINICAL TRIAL: NCT06473168
Title: Walking-related Mobility Assessment in Older People With Multimorbidity
Brief Title: Mobility Assessment in Multi-morbidity
Acronym: Multi-mobility
Status: Not yet recruiting | Type: Observational
Sponsor: Northumbria University (Other)
Collaborators: Newcastle University (Other)
Responsible Party: Principal Investigator, Ioannis Vogiatzis, Professor of Rehabilitation Sciences, Northumbria University
Other Study IDs: 700448
Record Dates: First submitted 2024-06-07; First posted 2024-06-25 (Actual); Last update posted 2024-06-25 (Actual); Status verified 2024-06

CONDITIONS: Arthritis; Asthma; Atrial Fibrillation; Bronchiectasis; Cancer; Chronic Kidney Diseases; Chronic Obstructive Pulmonary Disease; Coronary Heart Disease; Anxiety; Depression; Diabetes Mellitus; Heart Failure; Hypertension; Osteoporosis; Parkinson Disease; Peripheral Vascular Disease; Stroke; Transient Ischemic Attack
MeSH Terms: conditions — Arthritis; Asthma; Atrial Fibrillation; Bronchiectasis; Neoplasms; Renal Insufficiency, Chronic; Pulmonary Disease, Chronic Obstructive; Coronary Disease; Anxiety Disorders; Depression; Diabetes Mellitus; Heart Failure; Hypertension; Osteoporosis; Parkinson Disease; Peripheral Vascular Diseases; Stroke; Ischemic Attack, Transient

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Multimorbidity (the presence of two or more coexisting long-term conditions) is a significant challenge facing the NHS, especially given UK's ageing population and the association with high levels of illness burden and healthcare costs. Over 50% of adults >65 years have multiple long-term conditions (MLTCs).

Our group has validated a broad range of algorithms applied to single wearable sensors that have the potential to capture walking-related mobility outcomes (such as walking cadence and walking speed) accurately and reliably during activities of daily living across five single long-term conditions. These algorithms, however, cannot be readily applied to people with MLTCs because the effect of multimorbidity on mobility is amplified compared to single long-term conditions secondary to a greater number of complications and sequelae. Accordingly, the aim of this study is to validate algorithms that would allow robust estimation of walking-related mobility outcomes during daily life activities in MLTCs.

To meet our objectives, the investigators will perform: i) laboratory-based technical validation of existing and newly developed algorithms for walking-related mobility outcome detection; ii) unsupervised real-life validation of selected algorithms; and iii) examination of how well the validated walking-related mobility outcomes reflect global and disease specific characteristics in older adults with multimorbidity. The investigators will adopt an integrated patient-centric approach where patients with MLTCs will be engaged early in the project to provide input of their perception and concerns regarding mobility limitation in daily life activities.

The investigators aim to recruit 55 older adults (>65 years), men and women, with multiple long-term conditions with the following inclusion criteria: having two or more of the following conditions including osteoarthritis, rheumatoid arthritis, osteoporosis, type 2 diabetes, depression and/or anxiety, hypertension, coronary heart disease, heart failure, atrial fibrillation, chronic obstructive pulmonary disease, asthma, bronchiectasis, chronic kidney disease, cancer, or stroke within the last 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Adults ≥65 years old
* Able and willing to provide informed consent
* Able to read and write in English
* To be mobile (including the use of walking aids)
* Two or more of the following long terms conditions: Arthritis, Asthma, Atrial fibrillation, Bronchiectasis, Cancer, Chronic kidney disease, Chronic obstructive pulmonary disease, Coronary heart disease, Anxiety, Depression, Diabetes mellitus, Heart failure, Hypertension, Osteoporosis, Parkinson's disease, Peripheral vascular disease, Stroke or transient ischaemic attack

Exclusion Criteria:

* Unable to give consent for the study
* Severe mental health problems
* Active malignancy (on chemotherapy/radiotherapy/planned urgent surgery)

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patients will be recruited from outpatient clinics within the Newcastle upon Tyne Hospitals NHS Foundation Trust.
Sampling Method: Non-Probability Sample
Enrollment: 55 (Estimated)
Dates: Start 2024-12-01 (Estimated); Primary Completion 2025-10-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Cadence | 7-day real world assessment
  Walking cadence measured in the real world obtained from the Inertial Measurement Units placed on the lower back and the wrist measured in steps/minute.
Stride length | 7-day real world assessment
  Stride length measured in the real world obtained from the Inertial Measurement Units placed on the lower back and the wrist measured in meters.
Walking speed | 7-day real world assessment
  Walking speed measured in the real world obtained from the Inertial Measurement Units placed on the lower back and the wrist measured in m/s.
Stride duration | 7-day real world assessment
  Stride duration measured in the real world obtained from the Inertial Measurement Units placed on the lower back and the wrist measured in sec.

SECONDARY OUTCOMES:
Turning angle | 7-day real world assessment
  Measured in the real world obtained from the Inertial Measurement Unit placed on the lower back and the wrist expressed in deg/s.
Daily steps | 7-day real world assessment
  Measured in the real world obtained from the Inertial Measurement Unit placed on the lower back and the wrist expressed in steps/day.
Sedentarism | 7-day real world assessment
  Measured in the real world obtained from the Inertial Measurement Unit placed on the lower back and the wrist indicating time spent in different types of activities such as sitting down, lying, and walking expressed in minutes per day.

CONTACTS AND LOCATIONS:
Overall Officials: Laura Hutchinson, BSc, Study Chair — Northumbria University Newcastle